CLINICAL TRIAL: NCT00718835
Title: Incentive-based Smoking Cessation for Methadone Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Vermont Medical Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Stacey C. Sigmon, Associate Professor, University of Vermont Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01DA019550 (NIH); R01DA019550 (NIH)
Record Dates: First submitted 2008-07-17; First posted 2008-07-21 (Estimated); Last update posted 2014-02-21 (Estimated); Status verified 2014-02

CONDITIONS: Cigarette Smoking Among Patients Currently Receiving Methadone or Buprenorphine Treatment for Opioid Dependence
Keywords: smoking cessation; behavioral treatment; contingency management; opioid maintenance; methadone; buprenorphine
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Contingent Voucher condition (Active Comparator): Subjects in this condition will receive a brief education intervention plus voucher-based incentives contingent on demonstrating objective evidence of recent smoking abstinence.
  Interventions: Behavioral: incentive-based contingency management
- Noncontingent control condition (Placebo Comparator): Subjects assigned to this control condition will receive the brief education and vouchers delivered independent of smoking status and yoked to the schedule of voucher earnings in the Contingent Voucher condition.
  Interventions: Behavioral: incentive-based contingency management

INTERVENTIONS:
Behavioral: incentive-based contingency management — Direct comparison of Contingent versus Noncontingent incentives in promoting abstinence from smoking among opioid-treatment patients. The biochemical measures of breath carbon monoxide levels and urinary cotinine are used to confirm smoking status. Participants receive voucher-based incentives either contingent upon demonstrating abstinence from recent smoking (Contingent condition) or independent of smoking status (Noncontingent control condition).

SUMMARY:
The prevalence of cigarette smoking among patients receiving opioid agonist treatment, such as methadone or buprenorphine maintenance, is more than three-fold that of the general population and is associated with increased morbidity and mortality. The overarching goal of this project is to systematically develop a voucher-based contingency-management (CM) intervention for promoting initial and longer-term abstinence from cigarette smoking in patients receiving methadone or buprenorphine treatment for their opioid abuse.

DETAILED DESCRIPTION:
The prevalence of cigarette smoking among patients receiving opioid agonist treatment, such as methadone or buprenorphine maintenance, is more than three-fold that of the general population and is associated with increased morbidity and mortality. Despite these statistics, little is known about how to effectively help opioid-maintained patients to quit smoking. We believe a treatment that successfully promotes smoking cessation in these patients would offer exciting potential for dissemination. First, these treatment modalities are uniquely situated to offer an ideal setting for implementing smoking-cessation interventions. Many patients achieve significant periods of stability and drug abstinence and remain engaged in treatment for long periods of time, which can promote the frequent and prolonged clinical contact to enable success with smoking cessation. Second, opioid treatment programs often adhere to a uniform set of state and federal regulations, which could support the dissemination of an effective intervention throughout clinics across the country. Therefore, the overarching goal of this Behavior Therapy Development project is to systematically develop a voucher-based contingency-management (CM) intervention for promoting initial and longer-term abstinence from cigarette smoking in patients receiving methadone or buprenorphine treatment for their opioid abuse. Our first aim is to develop a CM treatment that will promote initial smoking abstinence in these patients using an intensive but brief 2-week intervention (Study 1). Our second aim will then be to integrate procedures for establishing initial abstinence with those designed for maintaining abstinence with the overarching goal of promoting smoking cessation that is sustained after the incentive program is discontinued (Study 2).

ELIGIBILITY:
Inclusion Criteria:

* For inclusion in the proposed study, subjects must report smoking 10 or more cigarettes per day and have smoked at least that amount for the past year. Subjects must be maintained on a stable methadone or buprenorphine dose for the month before study intake, with no evidence of regular illicit-drug abuse (<30% positive specimens for illicit drugs in the past 30 days).

Exclusion Criteria:

* Participants will be excluded if they are currently pregnant and/or nursing or if they report regular THC use and are unwilling to stop before beginning the study (THC use will confound CO values when we aim to monitor smoking status).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2007-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
percent of subjects abstinent during the second week of the two-week monitoring period | continuously and at end of 2-week trial

SECONDARY OUTCOMES:
mean days of continuous abstinence achieved during the 2-week abstinence monitoring period and mean number days abstinent (non-continuous) | continuously and at end of 2-week trial

CONTACTS AND LOCATIONS:
Overall Officials: Stacey C. Sigmon, Ph.D., Principal Investigator — University of Vermont, Department of Psychiatry
Locations (1):
- Substance Abuse Treatment Center, University of Vermont, Burlington, Vermont, United States

REFERENCES:
- [Derived] Sigmon SC, Miller ME, Meyer AC, Saulsgiver K, Badger GJ, Heil SH, Higgins ST. Financial incentives to promote extended smoking abstinence in opioid-maintained patients: a randomized trial. Addiction. 2016 May;111(5):903-12. doi: 10.1111/add.13264. Epub 2016 Jan 23. PMID 26638126